CLINICAL TRIAL: NCT03039829
Title: Short-Term Safety and Dose Effects of Different Forms of Creatine
Brief Title: Safety of Different Forms of Creatine
Acronym: NB9
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Nutrabolt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB2015-0684
Record Dates: First submitted 2017-01-20; First posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Nutritional Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Creatine nitrate, low dose (Experimental): Creatine nitrate at 3.0 grams (2.0 grams creatine; 1.0 gram nitrate, 3.0 grams dextrose)
  Interventions: Dietary Supplement: Creatine nitrate, low dose
- Creatine nitrate, high dose (Active Comparator): Creatine nitrate at 6.0 grams (4.0 grams creatine; 2.0 grams nitrate)
  Interventions: Dietary Supplement: Creatine nitrate, high dose
- Placebo (Placebo Comparator): Placebo at 6.0 grams dextrose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine nitrate, low dose — Creatine nitrate at 3.0 grams (2.0 grams creatine, 1.0 gram nitrate, 3.0 grams dextrose)
  Arms: Creatine nitrate, low dose
Dietary Supplement: Creatine nitrate, high dose — Creatine nitrate at 6.0 grams (4.0 grams creatine, 2.0 grams nitrate)
  Arms: Creatine nitrate, high dose
Dietary Supplement: Placebo — Placebo at 6.0 grams (6.0 grams dextrose)
  Arms: Placebo

SUMMARY:
This study will aim to determine whether ingesting creatine nitrate (CrN) at higher doses will differentially affect hemodynamic variables compared to a placebo.

DETAILED DESCRIPTION:
This study will examine the short-term (7 day) characteristics of ingesting creatine nitrate (CrN) compared to placebo on Chem-15 blood safety, heart rate, blood pressure, heart rate and blood pressure reactivity and self-reported side effects.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy
* At least 6 months immediate prior history of resistance training including bench press and leg press or squat

Exclusion Criteria:

* A history of treatment for metabolic disease (i.e., diabetes), hypertension, hypotension, thyroid disease, arrhythmias and/or cardiovascular disease
* Use of prescription medication (birth control is allowed)
* Pregnant or nursing or plan to become pregnant during the next month
* Creatine or nitrate use in the last eight weeks
* History of smoking
* History of drinking (i.e., 12 drinks per week or more)
* Use of nonsteroidal anti-inflammatory drugs (NSAIDs) including ibuprofen (Advil, Motrin, Nuprin, etc.), indomethacin (Indocin), naproxen (Aleve, Anaprox, Naprelan, Naprosyn), piroxicam (Feldene)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Measuring the blood pressure response to creatine nitrate ingestion | 7 days
Measuring the heart rate response to creatine nitrate ingestion | 7 days

SECONDARY OUTCOMES:
Measuring a blood chemistry panel 15 response to creatine nitrate ingestion | 7 days
Measuring the one Repetition Maximum (1 RM) muscle strength response to creatine nitrate ingestion | 7 days
Measuring the repetitions to failure muscle endurance response to creatine nitrate ingestion | 7 days
Measuring self-reported side effects of creatine nitrate ingestion | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University

IPD SHARING:
Plan to Share IPD: No